CLINICAL TRIAL: NCT03191617
Title: Nutrition of Premature Infants With Human Breastmilk Fortifier With Higher Protein Content and Long Chain Poli- Unsaturated Fatty Acids (LCPUFA)
Brief Title: Nutrition of Premature Infants With Human Breastmilk Fortifier
Acronym: EFORT-LM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NEOCOSUR (Other)
Responsible Party: Principal Investigator, Patricia Mena Nannig, MD, NEOCOSUR
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEOCOSUR
Record Dates: First submitted 2015-11-19; First posted 2017-06-19 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Growth Acceleration

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liquid human milk fortifier (Experimental): Liquid human milk fortifier which has higher protein content and also LCPUFA
  Interventions: Dietary Supplement: Human milk fortifier
- Powder human milk fortifier (Active Comparator): Powder human milk fortifier with less protein content and no LCPUFA
  Interventions: Dietary Supplement: Human milk fortifier

INTERVENTIONS:
Dietary Supplement: Human milk fortifier — Fortification of breastmilk with liquid human milk fortifier in premature infants
  Other Names: Mead Johnson´s Liquid Human Milk fortifier

SUMMARY:
The objective of the study is to compare two human milk fortifiers with different protein content and LCPUFA in a group of very low birth weight infants.

DETAILED DESCRIPTION:
This study is a multi-center, third party-blinded, randomized, controlled, parallel- group, prospective trial comparing growth with a liquid human milk fortifier with higher protein content and LCPUFA and a control powdered human milk fortifier added to breast milk and fed to premature infants. The trial will be conducted in 11 centers in Chile. The enrollment period is expected to be approximately 18 months. To allow for dropouts, approximately 160 participants will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Premature infant equal or under 31 weeks gestational age at birth
* Birth weight equal or under 1,250 g
* Predominantly fed breast milk (mother's milk or donor milk) on study day 0
* Appropriate birth weight for gestational age (AGA) - defined as birth weight between and inclusive of the 10th and 90th percentiles on the Fenton growth chart
* Singleton or twin birth (both twins do not need to qualify and be randomized into study)
* Birth weight is ≤1,000 g and participant is ≤ 40 days of age on study day 0
* Birth weight is above 1,000 g and participant is ≤ 30 days of age on study day 0
* Enteral intake of 80 mL/kg/d of unfortified breast milk on study day 0
* Anticipate mother's willingness to breast milk for at least 28 days from study day 0
* Signed informed consent obtained

Exclusion Criteria:

* History of underlying metabolic or chronic disease, congenital malformation, or any other condition which, in the opinion of the Investigator, is likely to interfere with: the ability of the participant to ingest food, normal growth and development of the participant, or the evaluation of the participant
* 5 minute APGAR score ≤ 4
* Major surgery that required general anesthesia prior to first day study (note: persistent ductus arterious ligation is allowed)
* Received pharmacologic doses of glucocorticoids during 3 consecutive days (72 hours) prior to or on day one of study (physiologic hydrocortisone administration up to 1.5 mg/kg/d is permitted)
* Ventilator-dependent and requiring ≥ 40% fraction of inspired oxygen (FiO2) on day one of study (ventilator dependent and requiring ≤ 40% FiO2 and/or nasal canula, and/or nasal continous positive airway pressure (CPAP) and/or oxygen hood is allowed)
* Grade III or IV bilateral intraventricular hemorrhage (IVH) prior to or on study day one
* Feeding intolerance to breast milk feedings on study day one
* Consumption of more than 3 feedings or 12 hours of continuous feeds of fortified breast milk prior to study day one
* Fluid restriction < 120 mL/kg/d
* History of creatinine >2.0 mg/dL 7 days prior to or on study day one
* Currently receiving or plan use of probiotics

Ages: 3 Days to 40 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Weight and linear growth | between entering study and 45 days in study or discharge, whatever first
  Weight increase in g/K/day and knee-to-heel length increase in mm/weeks, measured in one scale (+-5 g) and one kneenometer (special device to measure longitude) (+- 1mm) by one person for each center between entering study and 45 days in study or discharge

SECONDARY OUTCOMES:
Compare length of hospital- stay | days from the first day of study to discharge home , an average of 37 weeks of postconceptual age
  days from the first day of study to discharge home ( weight is one criteria for discharge)
Compare feeding tolerance | Between entering study and 45 days in study or discharge, if discharge first
  Daily record of residue, regurgitation and suspend of gastric feedings
Compare incidence of main preterm morbidities: necrotizing enterocolitis, bronchopulmonary dysplasia, retinopathy of prematurity and sepsis | Between entering study and 45 days in study or discharge, if discharge is first
  Incidence of necrotizing enterocolitis grade II or more, bronchopulmonary dysplasia as additional oxygen at 36 postconceptual weeks, retinopathy of prematurity with treatment and sepsis with positive hemoculture
Compare cost/benefits . The cost of use a fortificant and the benefit of growth velocity | Between entering study and 45 days in study or discharge, if discharge is first
  compare cost of total amount of fortifier used compare with cost of number of days of hospitalization, number of days in neonatal intensive care unit in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Mena, MD, Principal Investigator — Hospital Sotero Del Rio
Locations (1):
- Pontificia universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided